CLINICAL TRIAL: NCT04598659
Title: NHS England Proof of Concept - Smart Tech - Nene CCG
Brief Title: Nene Remote Monitoring Proof of Concept
Status: Completed | Type: Observational
Sponsor: Doccla UK (Industry)
Collaborators: NHS Nene Clinical Commissioning Group (Unknown); Northampton General Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Denis Shaughnessy, Chief Investigator, Doccla UK
Other Study IDs: NPoC1
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Cardiovascular Diseases; Respiratory Disease; Stroke
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Respiration Disorders; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This feasibility study is being conducted to investigate the practicalities and potential benefits of equipping patients with wearable monitoring devices.

DETAILED DESCRIPTION:
Vital signs are important indicators used in healthcare to inform a patient's treatment options and care plan. However, the opportunity to monitor vital signs is largely limited to the time a patient spends at a healthcare providers premises. This study is being conducted to see if the use of small wearable monitoring devices could help deliver a better service and improve patient care by continuing to monitor patients remotely.

The study is observational and has been designed to address two key questions:

1. Is it possible in principle to use the information captured from the devices to improve the treatment of the patient?
2. How practical is it to implement remote patient monitoring (RPM)?

To address these questions, consenting patients will be asked to wear a small adhesive biosensor for a short period of time following discharge from hospital (either as an outpatient or inpatient).

The data gathered by the device will be examined retrospectively and patients will not be monitored in real-time. Following the monitoring period, the vital signs data captured by the device will be analysed to see if it correlates with any unscheduled healthcare needs (such as unplanned GP appointments or emergency hospital visits). Specifically, the study team will be investigating whether the monitoring could have picked up a nascent problem before it became more serious, or whether monitoring could have saved the patient from having to make a trip to see their GP.

Information regarding the practicalities of implementing RPM will be captured by monitoring compliance and through an exit interview with participating patients.

ELIGIBILITY:
Inclusion Criteria:

* The participant is able to provide informed consent.
* The participant is able to comply with the English instructions for using a wearable device (e.g, follow simple instructions, able to answer the telephone, able to answer symptom questions, etc.).
* The participant may have been recently discharged from a hospital care setting (including emergency departments, ward and acute assessment units) to home (including a relative's home) or be currently admitted to a hospital care setting.
* The participant has a recent medical history that suggests there is a risk their health may deteriorate at home. In the first instance we will focus upon patients with at least one of the following conditions:
* Heart Failure (the patient being discharged),
* Arrhythmia (e.g. patient on the waitlist for a pacemaker)
* We will also consider patients with other conditions that present a risk of deterioration at home, for example: COPD, stable angina, liver failure, minor trauma, chronic kidney disease, stroke, hypertension, cancer ( e.g. recent surgery)

Exclusion Criteria:

* Patients that are clinically unstable (eg: respiratory distress, ongoing angina pectoris, sepsis, etc).
* Aphasia or other conditions that prevents the patient from adequately communicating with the researchers.
* Terminal diagnosis with life expectancy < 3 months.
* Ongoing renal dialysis, or other treatment that prevents the patient from being at home for extended periods.
* Dementia or uncontrolled psychiatric illness.
* Severe dermatitis or another skin disorder that prevents the patient from wearing a patch.
* Patient has a pacemaker or ICD
* Other inability, or unwillingness, to adequately co-operate with the RPM-team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who present themselves for care or consultation at the Northampton General Hospital during the period of the study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Patient compliance | 7 days (the monitoring period)
  The percentage of all participating patients for whom a complete and unbroken record of their vital signs is obtained throughout the duration of the agreed monitoring period.

SECONDARY OUTCOMES:
Device comfort assessed by a 5-point rating scale | 15 minutes
  Participants will be asked to rate how comfortable they found the device to wear during a telephone administered exit interview.
Convenience of remote monitoring assessed by a 5-point rating scale | 15 minutes
  Participants will be asked how the remote monitoring device affected their daily routine during a telephone administered exit interview. Responses will be collected using a 5-point rating scale of convenience.
The average time required to support patients through the remote monitoring process | 6 months
  The amount of time that the study team spends on-boarding patients (fitting the devices and explaining how they work) and supporting patients to use the devices will be recorded, to calculate the average time that staff will need to support each patient and estimate the resource requirement for implementing remote monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: David Sharman, Principal Investigator — Northampton General Hospital
Locations (1):
- Northampton General Hospital, Northampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No